CLINICAL TRIAL: NCT06416306
Title: Speech Intervention for Bilingual Children
Brief Title: Treatment Targets in Spanish and English Bilingual Speech Intervention
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Philip Combiths (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Sponsor-Investigator, Philip Combiths, Assistant Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 202109072; R21DC021249 (NIH)
Record Dates: First submitted 2024-05-07; First posted 2024-05-16 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Speech Sound Disorder
Keywords: speech; speech sound disorder; bilingual; treatment targets
MeSH Terms: conditions — Speech Sound Disorder; Speech

STUDY DESIGN:
Intervention Model Description: Two prospective treatment studies that share an identical study design, differing only in the language of treatment (Spanish or English). Both studies will employ a within- and across-subjects, single-subject experimental design (SSED) with multiple staggered baselines across two conditions (singleton consonant target vs. consonant cluster target).
Who Masked: Participant, Outcomes Assessor
Masking Description: Outcomes will be determined from phonetic transcription of participants' speech during assessment sessions. All transcriptions will be completed by research assistants unaware of the condition (simple or complex treatment target), arm of the study (English or Spanish language of intervention) or phase of the intervention study (Pre, Post, or Follow-up).
  The participant will be unaware of the relative complexity of their treatment target (i.e., condition: simple or complex).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Spanish Language Intervention (Experimental): Treatment will be conducted entirely in Spanish, targeting Spanish speech sounds. Treatment will follow a drill-play format.
  Interventions: Behavioral: Speech Intervention
- English Language Intervention (Experimental): Treatment will be conducted entirely in English, targeting English speech sounds. Treatment will follow a drill-play format.
  Interventions: Behavioral: Speech Intervention

INTERVENTIONS:
Behavioral: Speech Intervention — The treatment will begin with imitation, whereby the child will produce target words following the study clinician's verbal model with 1:1 clinician feedback for the accuracy of the child's productions. This will include explicit articulatory instruction (i.e., verbal and visual cues) to elicit correct target forms. When a child achieves 75% accuracy following a verbal model across 2 consecutive sessions or completes the 9th session (whichever is first), treatment will shift to spontaneous production, in which the child will produce target words spontaneously or through elicitation without a verbal model. Treatment materials will be images of treatment target words, interactive games and stories, and a standard set of toys.

SUMMARY:
The goal of this clinical trial is to learn which speech treatment targets result in the greatest amount of speech learning in Spanish-English bilingual children with speech sound disorders. The main questions it aims to answer are:

* Does linguistic complexity of the treatment target increase the amount of generalized learning within the treated language?
* Does linguistic complexity of the treatment target increase the amount of generalized speech across languages?

Researchers will compare intervention effects across treatment provided in English and Spanish to see if the effect differs according to the language of intervention.

Participants will:

* Attend between 12 and 18 45-minute speech intervention sessions in Spanish or English for up to 6 weeks
* Attend assessment visits before and after intervention
* Attend follow-up assessment visits 1 month and 2 months after intervention

DETAILED DESCRIPTION:
This study is a single-subject experimental design with staggered multiple baselines examining speech intervention for Spanish-English bilingual children with speech sound disorders. The study includes two arms based on the language of intervention (Spanish or English). Within each arm are two conditions that manipulate the linguistic complexity of the speech treatment target (simple consonant singleton or complex consonant cluster). Participants will be pseudo-randomly assigned to these arms and conditions.

The primary outcome is system-wide generalization; specifically, a) within-language and b) across-language generalization to untreated sounds. Accuracy data for the dependent variable will be derived from narrow phonetic transcription of participants' productions from speech probes in English and Spanish. The entire generalization probe is administered at each assessment visit (Pre, Post, and 1- and 2-Month Follow-Ups), and shorter subset probes targeting only monitored sounds are administered during Baselines and weekly during Treatment.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be regularly exposed to English for at least 3 months in one of the following ways: a) an English-speaking caregiver or sibling who interacts with the child on a daily basis in English, b) attendance at an English-speaking daycare, preschool, or elementary school.
* Caregivers will have reported concern with their child's speech development and/or reduced intelligibility on the Intelligibility in Context Scale in Spanish or English.
* Participants will present with 5 or more consonants or clusters missing from their phonetic inventories in each language to confirm presence of a speech sound disorder and sufficient gaps in phonological knowledge to warrant treatment.

Exclusion Criteria:

* Participants receiving speech or language treatment elsewhere during their participation in this project.

Ages: 3 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 16 (Estimated)
Dates: Start 2024-05-08 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Comprehensive Probe or Monitored Sounds Probe | At initial visit, 2-4 times across the 2 weeks prior to intervention, once per week during the 6-week intervention, within 1 week after intervention, 1 month after intervention, and 2 months after intervention
  Accuracy data for the dependent variable will be derived from narrow phonetic transcription of participants' productions from speech generalization probes in English and Spanish. Both protocols elicit ~300 word productions and sample each singleton consonant and consonant cluster in the respective language a minimum of three times in every permissible word position. The entire generalization probe is administered at each assessment visit (Pre, Post, and 1- and 2-Month Follow-Ups), and shorter subset probes targeting only monitored sounds are administered during Baselines and weekly during Treatment. All transcriptions will be completed by research assistants unaware of the condition (simple or complex treatment target), arm of the study (English or Spanish language of intervention) or phase of the intervention study (Pre, Post, or Follow-up).

CONTACTS AND LOCATIONS:
Locations (1):
- University of Iowa, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No